CLINICAL TRIAL: NCT05704439
Title: Cardiovascular Risk in Epilepsy: Pilot Feasibility and Efficacy Study of Neurologist-Initiated Treatment of Hypertension and Hyperlipidemia in an Underserved Minority Population in Los Angeles
Brief Title: Cardiovascular Risk Reduction in Epilepsy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not funded
Sponsor: University of California, Los Angeles (Other)
Collaborators: Olive View-UCLA Education & Research Institute (Other)
Responsible Party: Principal Investigator, Christopher Degiorgio, MD FAAN, Professor of Neurology in Residence, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CMD01
Record Dates: First submitted 2023-01-11; First posted 2023-01-30 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Epilepsy; Hypertension; Hyperlipidemia (E.G., Hypercholesterolemia)
Keywords: Epilepsy; Hyperlipidemia; Hypertension; Underserved
MeSH Terms: conditions — Epilepsy; Hypertension; Hyperlipidemias; Hypercholesterolemia | interventions — Antihypertensive Agents

STUDY DESIGN:
Intervention Model Description: Randomized Comparison of Neurologist initiated treatment of Hypertension or Hyperlipidemia versus usual care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Model 1-Neurologist Initiation of Treatment for Hypertension or Hyperlipidemia (Active Comparator): Neurologist Initiation of antihypertensive or treatment for hyperlipidemia
  Interventions: Drug: Neurologist Initiated Treatment
- Model 2-Usual Care (Placebo Comparator): Usual care
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Neurologist Initiated Treatment — Neurologist Initiated Treatment for Hypertension or Hyperlipidemia
  Other Names: antihypertensive agent or Hyperlipidemia agent
  Arms: Model 1-Neurologist Initiation of Treatment for Hypertension or Hyperlipidemia
Other: Placebo — Usual care
  Other Names: Usual Care
  Arms: Model 2-Usual Care

SUMMARY:
Epilepsy is a disabling and lethal neurological disease which affect 3.47 million Americans. Significant health care disparities exist in people with epilepsy (PWE). Hypertension and hyperlipidemia are highly prevalent and often go undertreated, and cardiovascular (CV) mortality is higher in people with epilepsy (PWE) than the general population. Preliminary data from our group shows that PWE have higher ACC-ASCVD risk scores than an age matched NHANES cohort without epilepsy. Preliminary data also demonstrate mortality rates in PWE due to hypertension, stroke, and diabetes are rising in the US, counter to the US general population.

This proposal seeks to test the feasibility, acceptability, and preliminary efficacy of a new care model for the underserved PWE in a public health setting. In this new model, neurologists guided by standardized treatment algorithms (ACC-ASCVD estimator+) propose and initiate pharmacological interventions for hypertension and hyperlipidemia.

DETAILED DESCRIPTION:
Epilepsy is a disabling and lethal neurological disease which affect 3.47 million Americans. Significant health care disparities exist in people with epilepsy (PWE). PWE are more likely to be Hispanic, Black, developmentally disabled and unemployed. Hypertension and hyperlipidemia are highly prevalent and often go undertreated, and cardiovascular (CV) mortality is higher in people with epilepsy (PWE) than the general population. Preliminary data from our group shows that PWE have higher ACC-ASCVD risk scores than an age matched NHANES cohort without epilepsy. Preliminary data also demonstrate mortality rates in PWE due to hypertension, stroke, and diabetes are rising in the US, counter to the US general population.

PWE on Medicaid, Medi-Cal and without insurance are more likely to experience delays to treatment and follow aberrant care pathways. Unexpected seizures and status epilepticus often result in transport to community and public health hospitals, where they are referred to neurology clinics, a process which may bypass primary care. As a result, PWE may have as their primary point of contact neurologists who traditionally do no monitor or treat hypertension or hyperlipidemia. This leads to gaps in care and missed opportunities to reduce CV risk.

This proposal seeks to test the feasibility, acceptability, and preliminary efficacy of a new care model for the underserved PWE in a public health setting. In this new model, neurologists guided by standardized treatment algorithms (ACC-ASCVD estimator+) propose and initiate pharmacological interventions for hypertension and hyperlipidemia.

We propose enrolling 150 subjects ages 40-79 with untreated or incompletely treated hypertension and/or hyperlipidemia. Subjects will be randomized 2:1 to Neurologist-initiated treatment (Model 1) versus usual care (Model 2). Subjects will be evaluated for blood pressure, blood chemistries, lipids, and HgA1C at baseline, one and three months. At 3-months, subjects randomized to usual care (Model 2) will be offered treatment if not yet initiated by primary care. If successful, results of this pilot study will provide needed feasibility and preliminary efficacy data for a large multicenter randomized trial of Neurologist initiated treatment of cardiovascular risk in the underserved with epilepsy

ELIGIBILITY:
Inclusion Criteria

* Epilepsy defined as G40.0-G40.9 in the electronic medical record, or seizure disorder prescribed at least one antiseizure medication
* Age 40-79 (age range defined by ACC-ASCVD risk estimator+)
* Untreated HTN defined as at least two sitting BPs > 130/80 in the last year prior to enrollment or on enrollment
* Hyperlipidemia defined as LDL > 70 mg/dl with 10-year ACC-ASCVD score > 7.5% or total LDL > 190, or ASCVD recommendation to initiate lipid lowering agent
* Intellectual Disability, developmental disorder or autism recorded in the electronic medical record (ICD-10 codes F70-F79, F84)

Exclusion Criteria:

* Stroke or cerebral hemorrhage < 1 year
* Documented poor compliance with treatment
* If intellectually disabled, if there is no caregiver to support or initiate therapy
* Pregnancy or person actively trying to become pregnant
* Blood Pressure > 180/110
* Known secondary cause of hypertension that causes concern regarding safety of the protocol.
* Arm circumference too large or small to allow accurate blood pressure measurement with available devices
* Diabetes mellitus,
* Glomerulonephritis treated with or likely to be treated with immunosuppressive therapy
* eGFR < 20 ml/min /1.73m2 or end-stage renal disease (ESRD)
* Cardiovascular event, procedure or hospitalization for unstable angina within last 3 months
* Symptomatic heart failure within the past 6 months
* A medical condition likely to limit survival to less than 3 years or a malignancy other than non-melanoma skin cancer within the last 2 years
* Any factors judged by the clinic team to be likely to limit adherence to interventions.
* Failure to obtain informed consent from participant
* Any organ transplant

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in ACC-ASCVD score from baseline | 3-months
  Percent change in ACC-ASCVD score (ACC-ASCVD) compared with baseline

SECONDARY OUTCOMES:
Systolic blood pressure | 3 months
  change in blood pressure (mmHg)
Total Cholesterol | 3 months
  change in total cholesterol (mg/dl) from baseline
LDL-low density lipoprotein | 3 months
  change in low density lipoprotein (mg/dl) from baseline
Compliance | 3 months
  Percent of enrolled subjects who complete visit three
Acceptability Rate | 3 months
  Rate: Number of medication proposals accepted by primary care physicians/number of medication proposals submitted to primary care physicians

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M DeGiorgio, MD, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No
pending